CLINICAL TRIAL: NCT04734353
Title: Efficacy, Safety and Tolerability of PrasugrEl 5mg or TIcagrelor 60mg in COmplex and Higher-Risk Indicated PCI/PatieNts: The Prospective, Randomized, Open-labeled, Blinded Endpoint (PROBE), Multi-center E5TION Trial
Brief Title: Prasugrel 5 mg vs. Ticagrelor 60 mg in CHIP (E5TION)
Acronym: E-5TION
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gyeongsang National University Hospital (Other)
Collaborators: U&I Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-5TION
Record Dates: First submitted 2020-08-18; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease
Keywords: High-risk coronary artery disease; Prasugrel; Ticagrelor
MeSH Terms: conditions — Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E5 group (Experimental): Escalation in CHIP
  Interventions: Drug: Prasugrel 5mg
- T60 group (Active Comparator): Escalation in CHIP
  Interventions: Drug: Ticagrelor 60mg

INTERVENTIONS:
Drug: Prasugrel 5mg — Prasugrel 20 mg loading, followed by prasugrel 5 mg/day for 12 months
  Other Names: Effient
  Arms: E5 group
Drug: Ticagrelor 60mg — Ticagrelor 120 mg loading, followed by ticagrelor 60 mg bid for 12 months
  Other Names: Brillinta
  Arms: T60 group

SUMMARY:
E5TION will evaluate the efficacy, safety and tolerability of tailored two regimens (prasugrel 5mg/d vs. ticagrelor 60mg bid) in high-risk patients undergoing PCI (CHIP: COmplex and Higher-Risk Indicated PCI/PatieNts).

DETAILED DESCRIPTION:
Because CHIP (COmplex and Higher-Risk Indicated PCI/PatieNts) has been related with the increased risk of ischemic events following PCI, there are unmet needs to develop the tailored strategies (e.g., intensified antiplatelet treatment) for this cohort. During antithrombotic treatment, East Asian patients have been prone to bleed compared with Western patients ("East Asian Paradox"). For example, standard-dose potent P2Y12 inhibitors (e.g., ticagrelor, prasugrel) vs. clopidogrel did not demonstrate the better net clinical benefit in patients with acute coronary syndrome. One of the tailored antiplatelet strategies for East Asian patients would be the de-escalated strategy of potent P2Y12 inhibitors (e.g., ticagrelor, prasugrel). The ISAR-REACT5 trial showed the lower ischemic event and better tolerability of ticagrelor vs. prasugrel in ACS patients. This E5TION trial will compare the efficacy, safety and tolerability of the de-escalated strategies (low-dose prasugrel and ticagrelor) in East Asian patients with CHIP character.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 and more; and
2. Subjects who scheduled for percutaneous coronary intervention(PCI) with Firehawk® drug-eluting stent
3. At least one of the following high-risk factors;

   * Clinical factors: diabetes, chronic kidney disease (GFR < 60ml/min/1.73m2), LV dysfunction (LV EF < 45%), or troponin (+).

     * Lesion- or procedure-related factors: left main PCI, chronic total occlusion, bifurcation lesion requiring two-stent technique, severe calcification, in-stent restenosis, multi-vessel PCI (≥ 2 vessels requiring stent implantation), PCI for ≥ 3 lesions, ≥ 3 stents implanted, or total stent length > 60 mm.

       * High platelet reactivity: VerifyNow PRU ≥ 266.

Exclusion Criteria:

1. Cardiogenic shock at the index admission
2. Bleeding tendency, congenital or acquired
3. Active bleeding or high-risk for major bleeding (e.g. active peptic ulcer disease, gastrointestinal pathology with a high-risk for bleeding, malignancies with a high-risk for bleeding)
4. Need for chronic oral anticoagulation
5. History of intracranial hemorrhage
6. Intracranial neoplasm, AV fistula or aneurysm
7. Platelet counts < 100,000/mm3
8. Liver cirrhosis with ascites or coagulopathy
9. Dialysis-impending or -dependent renal failure
10. Pregnant and/or lactating women
11. Increased risk of bradycardia events (sick sinus, AV block grade II or III, bradycardia-induced syncope)
12. Concomitant oral or i.v. therapy with strong CYP3A inhibitors (e.g., ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, grapefruit juice >1L/day), CYP3A substrates with narrow therapeutic indices (e.g., cyclosporine, quinidine), or strong CYP3A inducers (e.g., rifampin/ rifampicin, phenytoin, carbamazepine, dexamethason, phenobarbital) that cannot be safely discontinued
13. Concurrent medical condition with a life expectancy of less than 1 years

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-06-15 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Major bleeding and adherence to DAPT regimen | 1 year after PCI
  Incidence of major bleeding (BARC type 2, 3 or 5) and prevalence of discontinuation/switch of antiplatelet regimen

SECONDARY OUTCOMES:
MACE | 1 year after PCI
  Incidence of MACE (CV death, myocardial infarction, stent thrombosis, stroke or urgent revascularization)
Major bleeding | 1 year after PCI
  Incidence of BARC type 2, 3 or 5 bleeding
Major bleeding | 1 year post-PCI
  Incidence of ISTH major bleeding or clinically relevant non-major (CRNM) bleeding
Adherence to DAPT regimen | 1 year after PCI
  Prevalence of discontinuation/switch of antiplatelet regimen d/t side effect

OTHER OUTCOMES:
Platelet function test | 1 month after PCI
  VerifyNow PRU
Bleeding assessment | 1 month after PCI
  Assessment of BARC bleeding based on dedicated bleeding questionnaire
Dyspnea assessment | 1 month after PCI
  Assessment of dyspnea based on dedicated dyspnea questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoon Jeong, MD, PhD, Principal Investigator — Changwon Gyeongsang National University Hospital
Locations (8):
- South Korea (8):
  - Gyeongsang National University Changwon Hospital, Changwon, Gyeongsangnam-do
  - Gyeongsang National University Hospita, Jinju, Gyeongsangnam-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Kosin University Gospel Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital,, Busan
  - Inje University Busan Paik Hospital,, Busan
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schupke S, Neumann FJ, Menichelli M, Mayer K, Bernlochner I, Wohrle J, Richardt G, Liebetrau C, Witzenbichler B, Antoniucci D, Akin I, Bott-Flugel L, Fischer M, Landmesser U, Katus HA, Sibbing D, Seyfarth M, Janisch M, Boncompagni D, Hilz R, Rottbauer W, Okrojek R, Mollmann H, Hochholzer W, Migliorini A, Cassese S, Mollo P, Xhepa E, Kufner S, Strehle A, Leggewie S, Allali A, Ndrepepa G, Schuhlen H, Angiolillo DJ, Hamm CW, Hapfelmeier A, Tolg R, Trenk D, Schunkert H, Laugwitz KL, Kastrati A; ISAR-REACT 5 Trial Investigators. Ticagrelor or Prasugrel in Patients with Acute Coronary Syndromes. N Engl J Med. 2019 Oct 17;381(16):1524-1534. doi: 10.1056/NEJMoa1908973. Epub 2019 Sep 1. PMID 31475799